CLINICAL TRIAL: NCT06313554
Title: A Single-center, Single-arm, Open-label Clinical Study of Surufatinib Combined With Toripalimab and HAIC in Patients With Inoperable or Metastatic Intrahepatic Cholangiocarcinoma
Brief Title: Surufatinib Combined With Toripalimab and HAIC in the Treatment of Inoperable or Metastatic Intrahepatic Cholangiocarcinoma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Lu Wang, MD, PhD, Head of liver surgery department, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMPL-012-SH-ICC101
Record Dates: First submitted 2024-03-10; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Intrahepatic Cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Surufatinib Combined With Toripalimab and HAIC (Experimental): The first week dose of solantinib was 150mg, the second week and the subsequent cycle was 200 mg once a day (QD) orally, Q3W, and the drug was suspended for one day on the day of HAIC;
  Toripalimab: 240mg intravenous infusion d1, Q3W;
  HAIC: All patients received HAIC treatment on D1. Hepatic arterial perfusion therapy (HAIC) : a treatment cycle every 3 weeks for 4-6 consecutive cycles:
  Surufatinib and Toripalimab were administered continuously until intolerable toxicity, disease progression, withdrawal of informed consent, loss of follow-up, and investigator judgment that medication should be discontinued (whichever occurred first).
  Interventions: Drug: Surufatinib、Toripalimab、Gemcitabine、Oxaliplatin

INTERVENTIONS:
Drug: Surufatinib、Toripalimab、Gemcitabine、Oxaliplatin — The first week dose of Surufatinib was 150mg, the second week and the subsequent cycle was 200 mg once a day (QD) orally, Q3W, and the drug was suspended for one day on the day of HAIC; Toripalimab: 240mg intravenous infusion d1, Q3W;
  HAIC: All patients received HAIC treatment on D1. Hepatic arterial perfusion therapy (HAIC) : a treatment cycle every 3 weeks for 4-6 consecutive cycles:
  Surufatinib and Toripalimab were administered continuously until intolerable toxicity, disease progression, withdrawal of informed consent, loss of follow-up, and investigator judgment that medication should be discontinued (whichever occurred first).

SUMMARY:
This study is a single-arm, open-arm, single-center clinical study to explore the efficacy and safety of HAIC in combination with Surufatinib and Toripalimab in patients with inoperable or metastatic intrahepatic cholangiocarcinoma.

The study was divided into three stages: screening period, treatment period and follow-up period. During the treatment period, the tumor status was evaluated by imaging every 6 weeks (±7 days), and the efficacy was changed to every 8 weeks (±7 days) after 12 weeks until the disease progressed (RECIST 1.1) or death (during the treatment of the patient) or toxicity became intolerable. The tumor treatment status and survival status after the disease progression were recorded. Safety outcome measures included AE, changes in laboratory test values, vital signs and electrocardiogram changes.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects voluntarily joined the study and signed the informed consent, with good compliance and follow-up;
2. Inoperable or metastatic intrahepatic bile duct carcinoma confirmed by histopathology or cytology;
3. In accordance with the NCCN guidelines for intrahepatic cholangiocarcinoma diagnosis criteria, intrahepatic cholangiocarcinoma not suitable for radical resection was confirmed: R0 resection could not be obtained, liver was multiple, lymph node metastasis beyond the hepatic portal area and distant metastasis;
4. Male or female between the ages of 18 and 75 (including boundary values);
5. ECOG score: 0-1; Expected survival ≥12 weeks;
6. Liver function Child-Pugh grade A;
7. Have not received systematic treatment for inoperable or metastatic biliary tract cancer; Patients who had received adjuvant or neoadjuvant chemotherapy of one regimen and relapsed 6 months after the end of chemotherapy could be enrolled;
8. At least one measurable lesion (according to RECIST 1.1); Magnetic resonance imaging (MRI) enhancement or computed tomography (CT) enhancement were used to accurately measure the diameter of the lesion ≥1cm, and the study target lesion had not previously received local treatment (including but not limited to HIAC, radiofrequency ablation, argon helium knife, radiation therapy and other local treatments);
9. No serious organic diseases of heart, lung, brain and other organs;
10. The main organs and bone marrow functions are basically normal:

    1. Blood routine: white blood cells ≥ 4.0 x 109/L, neutrophils ≥ 1.5 x 109/L, platelets ≥ 80 x 109/L, hemoglobin ≥ 90g/L;
    2. International Standardized ratio (INR) and activated partial thromboplastin time (APTT) ≤1.5× upper limit of normal (ULN);
    3. Liver function: serum total bilirubin ≤ 2 x ULN; ALT/AST ≤ 2 x ULN; Serum albumin ≥28g/L;
    4. Renal function: serum creatinine ≤ 1.5 x ULN or eGFR≥60%, creatinine clearance (CCr) ≥60mL/min; To rule out urinary system infection, urine routine showed urine protein < 2+, ≥2+ patients should be collected 24 hours of urine protein volume < 1g;
    5. Normal cardiac function with left ventricular ejection fraction (LVEF)≥50% as measured by two-dimensional echocardiography;

Fertile male or female patients volunteered to use effective contraceptive methods, such as double barrier methods, condoms, oral or injectable contraceptives, and Iuds, during the study period and within 6 months of the last study medication. All female patients will be considered fertile unless they have undergone natural menopause, artificial menopause, or sterilization (such as hysterectomy, bilateral adnexectomy, or irradiation of radioactive ovaries).

Exclusion Criteria:

1. Participated in clinical trials of other anti-tumor drugs within 4 weeks before enrollment;
2. Patients with a history of TACE treatment and who had previously received any immune or targeted therapy were excluded; Patients with a history of hepatectomy, postoperative recurrence, and no systemic therapy were included
3. The investigators determined that liver metastases accounted for 90% or more of the total liver volume;
4. Patients who have previously received an organ transplant or are planning an organ transplant;
5. Patients with obstructive jaundice but yellowing is not as expected;
6. Have had other malignancies within the past 5 years, except basal cell or squamous cell carcinoma of the skin after radical surgery, or carcinoma in situ of the cervix;
7. Patients who have had or are currently having any brain metastases;
8. Other strong inducers or suppressors of CYP3A4 were taken within 2 weeks prior to the first study;
9. Received any surgery (except biopsy) or invasive treatment or operation within 4 weeks before enrollment, and the surgical incision was not completely healed (except intravenous catheterization, puncture drainage, etc.);
10. Electrolyte abnormalities identified by the investigator as clinically significant;
11. The patient currently has medically uncontrolled hypertension, defined as: systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg;
12. Urine routine indicated urinary protein ≥2+, and 24-hour urinary protein volume > 1.0g;
13. Patients whose tumors are judged by the investigators to be at high risk of invading vital blood vessels and causing fatal massive bleeding during the follow-up study;
14. Patients with evidence or history of significant bleeding tendency within 3 months prior to enrollment (bleeding within 3 months > 30 mL, hematemesis, stool, stool blood), hemoptysis (within 4 weeks > 5 mL fresh blood); People with a history of inherited or acquired bleeding or coagulation disorders. There were clinically significant bleeding symptoms or definite bleeding tendencies within 3 months prior to enrollment, such as gastrointestinal bleeding and hemorrhagic gastric ulcer;
15. Clinically significant cardiovascular disease, including but not limited to acute myocardial infarction, severe/unstable angina pectoris, or coronary artery bypass grafting within 6 months prior to enrollment; New York Heart Association (NYHA) Grades for Congestive Heart Failure > Level 2; Ventricular arrhythmias requiring medical treatment; Electrocardiogram (ECG) showed QT c interval ≥480 ms;
16. Active or uncontrolled severe infection (≥CTCAE grade 2 infection);
17. Unmitigated toxicity higher than CTCAE grade 2 due to any previous anticancer therapy, excluding alopecia, lymphocytopenia, and oxaliplatin grade ≤2 neurotoxicity;
18. Women who are pregnant (positive pregnancy test before medication) or breastfeeding;
19. Any other medical condition, clinically significant metabolic abnormality, physical abnormality or laboratory abnormality, which, in the investigator's judgment, reasonably suspects that the patient has a medical condition or condition that is not suitable for the use of the investigational drug (such as having seizures and requiring treatment), or which would affect the interpretation of the study results or place the patient at high risk;
20. Known human immunodeficiency virus (HIV) infection; Known history of clinically significant liver disease, including viral hepatitis [Known hepatitis B virus (HBV) carriers must rule out active HBV infection, i.e., positive HBV DNA (>1×104 copies /mL or > 2000 IU/ml); known hepatitis C virus infection (HCV) and HCV RNA positive (>1×103 copies /mL), or other hepatitis, cirrhosis;
21. The presence of any active, known or suspected autoimmune disease (including but not limited to: myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, enteritis, multiple sclerosis, vasculitis, glomerulonephritis, uveitis, pituitaritis, hyperthyroidism, etc.);
22. Known allergic reactions to other monoclonal antibodies or to any component of solvatinib;

According to the investigators' judgment, the patients had other factors that might affect the study results or lead to the forced termination of the study, such as alcoholism, drug abuse, other serious diseases (including mental illness) requiring combined treatment, serious laboratory abnormalities, and family or social factors that would affect the safety of the patients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2024-05-20 (Estimated); Primary Completion 2024-05-20 (Estimated); Study Completion 2027-05-20 (Estimated)

PRIMARY OUTCOMES:
ORR objective response rate | 24 months
  objective response rate (ORR)Defined as percentage of participants achieving assessed complete response (CR) and partial response (PR) by the investigator according to the RECIST 1.1.

SECONDARY OUTCOMES:
Progression-Free Survival(PFS) | 24 months
  PFS is defined as the time from enrollment to the first documented disease progression or death due to any cause, whichever occurs first.Responses are according to the Response Evaluation Criteria in Solid Tumors version 1.1(RECIST 1.1) as assessed by investigator
OS overall survival | 24 months
  OS is the time from enrollment to death due to any cause.
DCR disease control rate | 24 months
  DCR was defined as the percentage of participants who have a confirmed complete response (CR)or partial response (PR)or stable disease (SD) per RECIST 1.1 as assessed by investigator
Adverse events as assessed by NCI CTCAE v5.0 | 24 months
  overall incidence of adverse events (AE); incidence of grade 3 or higher AE; incidence of severe adverse events (SAE); incidence of AEs leading to discontinuation of drug use; incidence of AEs leading to suspension of drug use

IPD SHARING:
Plan to Share IPD: No